CLINICAL TRIAL: NCT05821140
Title: Evolution of the Maturation of Orofacial Functions and of the Masticatory Function During a Rehabilitation Program, in Children With Different Types of Deterioration in Oral Health
Brief Title: Orofacial Functions and Masticatory Function in Children With Different Types of Deterioration in Oral Health
Acronym: KIDYCROC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Odontologie Clinique UR4847 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2021 COLLADO; 2021-A00478-33 (Other: 2021-A00478-33)
Record Dates: First submitted 2022-12-09; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-11

CONDITIONS: Mastication; Disability; Oral Stage; Child Development
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- children with ECC (Experimental): Children under 6 with early childhood caries receiving comprehensive dental treatment under general anesthesia
  Interventions: Procedure: dental treatment for global oral rehabilitation; Other: oral health check up
- Children with orofacial dysmorphologies/malocclusion (Experimental): Children with orofacial dysmorphologies/malocclusion associated or not with a general condition and in need of a functional or orthodontic treatment
  Interventions: Procedure: dental treatment for global oral rehabilitation; Other: oral health check up
- Children with dental abnormalities (Experimental): Children with dental abnormalities associated or not with a general condition and in need of conservative, orthodontic or prosthetic treatment
  Interventions: Procedure: dental treatment for global oral rehabilitation; Other: oral health check up
- children with healthy oral state (Experimental): children with healthy oral state in the course of their annual follow-up visits.
  Interventions: Other: oral health check up

INTERVENTIONS:
Procedure: dental treatment for global oral rehabilitation — dental treatment can include conservative, orthodontic, prosthetic or surgical procedures
  Arms: Children with dental abnormalities; Children with orofacial dysmorphologies/malocclusion; children with ECC
Other: oral health check up — regular preventive follow-up visit (every 6 months)

SUMMARY:
This project aims at studying the evolution of masticatory function (food bolus granulometry, masticatory behavior, muscle activity and masticatory performance) during oral rehabilitation, in children with different types of oral health impairment.

Secondary objectives are to study the relationships between children masticatory function (food bolus granulometry, masticatory behavior, muscle activity and masticatory performance) and its evolution during oral rehabilitation, and:

* their type of oral health alteration
* their eating behaviors
* their height and weight status

During examination the following parameters are collected:

* Various clinical indicators of oral health
* The child's weight and height
* Frequency and nature of orofacial dysfunctions
* The oral health related quality of life of children and their families
* Chewing tests are performed (chewing gum, natural food such as carrot, cereals, and cheese samples, samples of gelatins of different hardness)

Examination and differents tests are performed every six months for a total of 5 years (per participant)

The dental care procedures performed during the study were carried out in the usual way.

DETAILED DESCRIPTION:
This project aims at studying the masticatory parameters and their evolution in children receiving oral rehabilitation at the special care unit (Odontology Department, CHU Estaing, Clermont-Ferrand), for different types of oral health alterations. These data could be used to support the validity of procedural guidelines in the field of functional rehabilitation in pediatric dentistry. The impact of the type of oral alteration on mastication, and the influence of the masticatory function on the quality of life, the eating habits and the height and weight status of children will also be analyzed.

The main objective is to study the evolution of masticatory function (food bolus granulometry, behavior, muscle activity and performance) during a rehabilitation program, in children with different types of oral health impairment.

Secondary objectives are to study the relationships between children masticatory function (food bolus granulometry, masticatory behavior, muscle activity and masticatory performance) and its evolution during oral rehabilitation, and:

* their type of oral health alteration
* their eating behaviors
* their height and weight status

This is a follow-up study using criteria from clinical orofacial examination, questionnaires, video recordings of natural food chewing sequences and analysis of food bolus.

Indeed, objective and non-invasive indicators of oro-facial functions and mastication are recorded as part of the usual follow-up of children (according to the recommendations of the American Association of Pediatric Dentistry 2020) during observations (live or on video recordings outside the presence of the family) or interviews with the child and his/her parents (questionnaires), or following masticatory tests.

During children examination, and after questionnaires are completed with the parents or the child himself, these data are collected:

* Various clinical indicators of oral health (caod/CAOD; PUFA; ICDAS)
* The child's weight and height for the calculation of the Body Mass Index (BMI) as a clinical indicator of the child's growth
* Frequency of orofacial dysfunctions (NOT-S test)
* The impact of oral health on the quality of life of children and their families (ECOHIS or COHIP tests depending on age)

The following parameters are collected from chewing tests:

* Children's chewing behavior described by the family (feeding behaviors) or observed during the visit (clinical index of "quality of muscle function during chewing") or determined outside the presence of the family from video recordings made during the visit while chewing test foods (chewing kinematic parameters).
* Granulometry of natural food boluses (D50: median particle size of food boluses)
* A chewing performance measured by the heterogeneity of a two-colored chewing gum after chewing for a defined number of cycles.
* The muscular activity during mastication of samples of gelatins of different hardness, carried out with recording of the masseter and temporal muscles activity (EMG)

The dental care procedures performed during the study were carried out in the usual way.

Examination and differents tests are performed every six months for a total of 5 years (per participant).

ELIGIBILITY:
Inclusion Criteria:

* All children, from 3 to 17 years old (inclusion limits), attending the special dental care unit of the CHU Estaing in Clermont Ferrand or the CH Guy Thomas in Riom are included in the study:
* Children and adolescents who have given their consent (6-17 years) and whose legal guardians have given their consent.
* Children (3-6 years old) with consent from the legal guardian.
* The subject is affiliated with a Social Security system.

This may include:

1. children with multiple caries, requiring full rehabilitation under sedation or general anesthesia +/- prosthetic rehabilitation,
2. children with orofacial dysmorphologies/malocclusions, associated or not with a general syndrome, requiring orthodontic and/or prosthetic treatment
3. children with dental abnormalities, associated or not with a general syndrome, requiring conservative, orthodontic and/or prosthetic treatment,
4. children with a healthy oral status in the course of their bi-annual oral health chek-up.

Exclusion criteria:

* Children with an ASA III or IV category according to the American Society of Anesthesiologists
* Children who do not have a solid diet due to severe neuromotor disorders.
* Children for whom a geographical or organizational barrier prevents follow-up in the service, children in social placement
* Children over 18 years of age
* Children (6-17 years) who do not volunteer to participate
* Children (6-17 years old) who are unable to give consent to participate in the research.
* Children for whom one of the legal guardians refuses to participate in the study
* Children whose legal guardians are not capable of giving informed consent.
* Children who are not affiliated to a Social Security system.
* Pregnant or nursing teenagers

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Particle size analysis of ready to swallow natural food bolus | at 6 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 12 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 18 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 24 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 36 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 48 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.
Particle size analysis of ready to swallow natural food bolus | at 60 months
  Particle size analysis (D50) of ready to swallow natural food boluses of carrot, cheese, or cereals.

SECONDARY OUTCOMES:
Correlation between mastication capability, and the type of oral health alteration | every 6 months for 1year, and then each year for 4 years
  Mastication capability is evaluated by particle size analysis (D50).
  The type of oral health alterations are defined by
  * presence of multiple caries
  * oro facial dysmorphologies
  * dental abnormalities
  * health oral state
Correlation between mastication behavior and the type of oral health alteration | every 6 months for 1year, and then each year for 4 years
  Mastication behavior is measured by measuring the number of food refusals during mastication tests, measuring the kinematic parameters (number of cycle (nc), mastication time (T) to calculate the masticatory frequency (nc/T)
  The type of oral health alterations are defined by
  * presence of multiple caries
  * oro facial dysmorphologies
  * dental abnormalities
  * health oral state
Correlation between mastication performance and the type of oral health alteration | every 6 months for 1year, and then each year for 4 years
  Mastication performance is evaluated by measuring the heterogeneity of the color of a bicolor chewing gum masticated during a given number of cycles (chewgum test) (Hue standard deviation)
  The type of oral health alterations are defined by
  * presence of multiple caries
  * oro facial dysmorphologies
  * dental abnormalities
  * health oral state
Correlation between muscle activity and the type of oral health alteration | every 6 months for 1year, and then each year for 4 years
  Muscle activity will be evaluated by measuring the electromyographic activity of masseter and temporal muscles during mastication of gelatines of various hardness.
  The type of oral health alterations are defined by
  * presence of multiple caries
  * oro facial dysmorphologies
  * dental abnormalities
  * health oral state
Correlation between mastiaction capability and quality of life | every 6 months for 1year, and then each year for 4 years
  The quality of life will be assessed using questionnaires:
  * ECOHIS for children less than 6 years old
  * COHIP for children above 6 years old
  Mastication capability is evaluated by particle size analysis (D50).
Correlation between mastication behavior and quality of life | every 6 months for 1year, and then each year for 4 years
  The quality of life will be assessed using questionnaires:
  * ECOHIS for children less than 6 years old
  * COHIP for children above 6 years old
  Mastication behavior is measured by measuring the number of food refusals during mastication tests, measuring the kinematic parameters (number of cycle (nc), mastication time (T) to calculate the masticatory frequency (nc/T)
Correlation between mastication muscular activity and quality of life | every 6 months for 1year, and then each year for 4 years
  The quality of life will be assessed using questionnaires:
  * ECOHIS for children less than 6 years old
  * COHIP for children above 6 years old
  Muscle activity will be evaluated by measuring the electromyographic activity of masseter and temporal muscles during mastication of gelatines of various hardness.
Correlation between mastication performance and quality of life | every 6 months for 1year, and then each year for 4 years
  The quality of life will be assessed using questionnaires:
  * ECOHIS for children less than 6 years old
  * COHIP for children above 6 years old
  Mastication performance is evaluated by measuring the heterogeneity of the color of a bicolor chewing gum masticated during a given number of cycles (chewgum test) (Hue standard deviation)
Correlation between mastication capability and eating habits | every 6 months for 1year, and then each year for 4 years
  Eating habits are measured by measuring the number of food refusals and texture adaptation at home according to the 7 categories of food (PNNS)
  Mastication capability is evaluated by particle size analysis (D50).
Correlation between mastication behavior and eating habits | every 6 months for 1year, and then each year for 4 years
  Eating habits are measured by measuring the number of food refusals and texture adaptation at home according to the 7 categories of food (PNNS)
  Mastication behavior is measured by measuring the number of food refusals during mastication tests, measuring the kinematic parameters (number of cycle (nc), mastication time (T) to calculate the masticatory frequency (nc/T)
Correlation between muscular activity and eating habits | every 6 months for 1year, and then each year for 4 years
  Eating habits are measured by measuring the number of food refusals and texture adaptation at home according to the 7 categories of food (PNNS)
  Muscle activity will be evaluated by measuring the electromyographic activity of masseter and temporal muscles during mastication of gelatines of various hardness.
Correlation between mastication performance and eating habits | every 6 months for 1year, and then each year for 4 years
  Eating habits are measured by measuring the number of food refusals and texture adaptation at home according to the 7 categories of food (PNNS)
  Mastication performance is evaluated by measuring the heterogeneity of the color of a bicolor chewing gum masticated during a given number of cycles (chewgum test) (Hue standard deviation)
Correlation between mastication behavior and height and weight status | every 6 months for 1year, and then each year for 4 years
  Mastication behavior is measured by measuring the number of food refusals during mastication tests, measuring the kinematic parameters (number of cycle (nc), mastication time (T) to calculate the masticatory frequency (nc/T)
  Height and weight status is evaluated by calculating the BMI (body mass index) of children
Correlation between muscular activity and height and weight status | every 6 months for 1year, and then each year for 4 years
  Muscle activity will be evaluated by measuring the electromyographic activity of masseter and temporal muscles during mastication of gelatines of various hardness.
  Height and weight status is evaluated by calculating the BMI (body mass index) of children
Correlation between mastication performance and height and weight status | every 6 months for 1year, and then each year for 4 years
  Mastication performance is evaluated by measuring the heterogeneity of the color of a bicolor chewing gum masticated during a given number of cycles (chewgum test) (Hue standard deviation)
  Height and weight status is evaluated by calculating the BMI (body mass index) of children

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Collado, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No